CLINICAL TRIAL: NCT04383301
Title: Combined Corneal Wavefront-guided Transepithelial Photorefractive Keratectomy and Accelerated Corneal Collagen Cross-linking Following Intra Corneal Ring Segment Implantation in Management of Moderate Keratoconus
Brief Title: Combined Corneal Wavefront-guided TPRK and ACXL Following ICRS Implantation in Management of Moderate Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaaban Elwan (Other)
Responsible Party: Sponsor-Investigator, Shaaban Elwan, Assistant professor of ophthalmology, Minia University
Organization: Minia University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Minia University & SFH-2
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Intervention Model Description: Intracorneal ring segment (ICRS) followed by accelerated corneal cross linking (ACXL) and wafe front guided transepithelial photorefractive keratotomy (TPRK)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra corneal ring segment (Active Comparator): Intra corneal ring segment implantation for moderate keratoconus patients
  Interventions: Procedure: Intracorneal ring segment implantaion as the first stage
- Corneal Wavefront-guided TPRK and ACXL (Active Comparator): Combined Corneal Wavefront-guided Transepithelial Photorefractive Keratectomy and Accelerated Corneal Collagen Cross-linking following intracorneal ring segment by at least three months
  Interventions: Procedure: ACXL and wafe front guieded TPRK as the second stage

INTERVENTIONS:
Procedure: Intracorneal ring segment implantaion as the first stage — Intracorneal ring segment (ICRS)
  Other Names: ICRS
  Arms: Intra corneal ring segment
Procedure: ACXL and wafe front guieded TPRK as the second stage — Accelerated corneal cross linking (ACXL) and wafe front guided transepithelial photorefractive keratotomy (TPRK)
  Other Names: ACXL and TPRK
  Arms: Corneal Wavefront-guided TPRK and ACXL

SUMMARY:
Background: Keratoconus leads to gradual progressive loss of vision in young and adult patients. For visual rehabilitation and to hinder keratoconus progressionthe investigators designed this study to help the keratoconus patients to improve and stabilize their vision.

Design: This is a prospective consecutive uncontrolled study.

Patients and Methods:

This study includes 36 eyes of 36 patients with moderate degree o keratoconus (KC) undergoing combined wave front guided transepithelial photorefractive keratectomy (TPRK) and accelerated corneal collagen crosslinking (ACXL) after intracorneal ring segment (ICRS) implantation. Uncorrected distance visual acuity (UDVA), corrected distance visual acuity (CDVA), manifest refraction spherical equivalent (MRSE), corneal indices based on Scheimpflug tomography, higher-order aberrations (HOAs) will be evaluated at baseline, after ICRS implantation, and at1, 3, 6, and 12 months after combined TPRK and CXL.

DETAILED DESCRIPTION:
Patients and Methods:

This study conducted upon 36 eyes of 36 patients with moderate keratoconus who undergoing combined corneal wavefront-guided TPRK and accelerated corneal CXL at least 3 months after ICRS implantation in the period between October, 2018 and April 2020, at the Security Forces Hospital, Ophthalmology Department, Riyadh, Kingdom of Saudi Arabia. The study was approved by SFHP ethical board committee (IRB registraion number: 18-289-54) and was adhered to the tenets of the Declaration of Helsinki as well as followed good clinical practices. All patients provided informed written consent for the study and for publication. All included patients undergoing combined corneal wavefront guided TPRK and corneal ACXL at least 3 months after ICRS implantation. Grading of keratoconus was based on the Amsler Krumeich classification. Progression was defined as one or more of the following changes over a period of 6 months: an increase of ≥1.00 diopter (D) in maximal keratometry values, an increase of ≥1.00 D in manifest cylinder, and an increase of ≥ 0.50 D in MRSE.

Examinations and measurements:- At baseline, the preoperative examination included UDVA, CDVA, manifest and cycloplegic refraction, slit lamp biomicroscopy, tonometry, Pentacam camera, tomography, and dilated fundus examination using binocular ophthalmoscopy. If patient use contact lenses it should be stopped 3 weeks before exam date, and medical history, including any systemic diseases, were recorded. After ICRS implantation (before combined TPRK and ACXL), and at 1, 3, 6, and 12 months after combined TPRK and CXL, all patients undergoing complete ophthalmic examinations, which included examinations for UDVA and CDVA with a Snellen chart, manifest refraction (MR). The corneal indices measured at the 8-mm zone using the Scheimpflug tomography system with Pentacam camera (OCULUS- Netzteil Art., Pentacam HR, Germany), and for measuring changes in corneal aberrations, including HOAs, coma, and spherical aberrations, corneal wavefront analysis implemented using corneal topographic data with tomography (Sirius, SCHWIND eye-tech-solutions GmbH, Kleinostheim, Germany). Root mean square (RMS) values of the corneal HOAs, with analysis up to the 7th order by expanding the set of Zernike polynomials, were calculated. Any postoperative complications, corneal haze , wound healing time were estimated. Patients overall satisfaction for the procedure were asked at last follow up and all data were recorded.

Surgical technique:-

First step procedure:

Before the surgery, tetracaine hydrochloride 0.5% ophthalmic solution (Bausch & Lomb, Minims) and moxifloxacin 0.5% (Vigamox, Alcon Co.) drops were instilled 3 times within a 5-minutes interval. The eyelids were prepared with antiseptic Chlorohexidine Gluconate 0.05% solution (Saudi Medical Solution Company). All patients undergoing femtosecond laser enabled ICRS implantation. An Intacs SK intra-corneal ring (6.0 mm optical zone; fixed arc length of 150∘; angulation 30∘) was implanted in the cornea. The ring segment thickness sizes were decided according to the nomogram provided by the manufacturer. The incision was placed at the steepest meridian and the depth of the ring tunel was set at 75-80% of the thinnest pachymetry reading. After surgery, a bandage contact lens (BIOMEDICS Evolution CL ocufilcon D 45%, water 55%) was placed to be removed after incision healing. Postoperative use of moxifloxacin 0.5% (Vigamox, Alcon Co.) eye drops 4 times/ day for two weeks, tobradex eye drops (Tobramycin 0.3%- dexamethasone 0.1%, Alcon Co.) with tapering dose for 1 month, and sodium hyaluronate 0.2% ( Hyfresh eye drops, Jamjoom Pharma Co.) eye drops QID for 3 months.

Second step procedure:

After at least 3 months with average 3.9 ± 2.2 and range (3-5) months from the ICRS implantation and when the mean keratometry stabilized and not decreased > 1 diopter from the previous visit, all patients were scheduled for combined corneal wavefront-guided TPRK and accelerated CXL. TPRK between the corneal ring segments were performed using Amaris excimer LASER 193 nm, version 750 S (Schwind eye-tech-solutions GmbH& Co. KG, Mainparkstrasse, Kleinostheim, Germany. The ablation profile was planned using the integrated Optimized Refractive Keratectomy-Custom Ablation Manager software (Schwind eye-tech-solutions GmbH and Co KG). Using this software, ablation was planned based on clinical parameters, including manifest refraction, pachymetry, and corneal wavefront data (up to the 7th order aberrations) and topography obtained with the Sirius topographer. The maximum ablation depth was limited to ( 50- 60 micro m), and then mitomycin C 0.02% (MMC) was applied for 20 seconds to reduce postoperative haze followed by eye irrigation with balanced saline solution (BSS). Riboflavin 0.1 % with hydroxypropyl methylcellulose (Vibex Rapid; Avedro Inc., Waltham, MA, USA) is soaked onto the corneal surface for 10 minutes immediately after excimer laser ablation. Riboflavin solution were added at 2 minutes interval during the soaking process after which the eye was irrigated with cold BSS. After completion of soaking, Ultra viollet A exposure (wavelength: 365 nm) was performed for 10 minutes at an irradiance of 9 mW/cm², to give a total radiant exposure of 5.4 J/cm² and intermittent riboflavin drops application during radiant exposure.

At the end of the surgery a bandage contact lens was placed, and the same previous postoperative medications were used beside pain keller oral tablet was perscribed if needed.

Statistical Analysis:- The investigators recorded all patients' data in Microsoft Excel Sheet, then copied and analyzed using A Graph Pad Prism 8 program; Paired student's t-test was used for the UDVA & CDVA means in log MAR values and for MRSE means. One way ANOVA was used for corneal indices. For all tests, a (P value < 0.05) was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with age > 20 years old and intolerant to contact lense use
* patients had moderate keratoconus (45-54 D in both meridians) without corneal scarring
* Central pachymetry ≥ 400 μm and if progression had been noted over the previous 6 months.

Exclusion Criteria:

* Patients with central or paracentral corneal scarring
* Central pachymetry <400 μm, systemic autoimmune disease
* History of herpetic keratitis, pregnancy, lactation, or severe dry eye syndrome.

Ages: 20 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
UDVA | one year
  Uncorrected distance visual acuity
CDVA | one year
  corrected distance visual acuity
Refractive changes | one year
  Refractive changes in the mean sphere, mean cylinder and manifest refractive spherical equivalent (MRSE)
Corneal Indices | 0ne year
  All corneal indices including steep, flat, mean and maximal keratometries

SECONDARY OUTCOMES:
HOA and coma aberrations | 1 year
  final root mean square (RMS) high orders aberrations (HOAs) and coma aberrations from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf M Bakhsh, MD, Principal Investigator — Security Forces Hospital Program
Locations (1):
- Security forces hospital, Riyadh, Central, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Tuwairqi WS, Osuagwu UL, Razzouk H, Ogbuehi KC. One-Year Clinical Outcomes of a Two-Step Surgical Management for Keratoconus-Topography-Guided Photorefractive Keratectomy/Cross-Linking After Intrastromal Corneal Ring Implantation. Eye Contact Lens. 2015 Nov;41(6):359-66. doi: 10.1097/ICL.0000000000000135. PMID 25839343
- [Background] Lee H, Kang DSY, Ha BJ, Choi JY, Kim EK, Seo KY, Kim TI. Visual rehabilitation in moderate keratoconus: combined corneal wavefront-guided transepithelial photorefractive keratectomy and high-fluence accelerated corneal collagen cross-linking after intracorneal ring segment implantation. BMC Ophthalmol. 2017 Dec 29;17(1):270. doi: 10.1186/s12886-017-0666-1. PMID 29284455
- [Background] Koh IH, Seo KY, Park SB, Yang H, Kim I, Kim JS, Hwang DG, Nam SM. One-Year Efficacy and Safety of Combined Photorefractive Keratectomy and Accelerated Corneal Collagen Cross-Linking after Intacs SK Intracorneal Ring Segment Implantation in Moderate Keratoconus. Biomed Res Int. 2019 Jul 8;2019:7850216. doi: 10.1155/2019/7850216. eCollection 2019. PMID 31360724